CLINICAL TRIAL: NCT02653118
Title: A Registry-Based Extension of Protocol V503-001 in Countries With Centralized Cervical Cancer Screening Infrastructures to Evaluate the Long-Term Effectiveness, Immunogenicity, and Safety of Multivalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine as Administered to 16- to 26- Year-Old Women
Brief Title: Long-term Follow-up of Broad Spectrum Human Papillomavirus (HPV) Vaccine Study in Women (V503-021)
Status: Active, not recruiting | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: V503-021; 2013-003549-40 (EudraCT Number)
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cervical Cancer; Vulvar Cancer; Vaginal Cancer; Genital Warts; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata; Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: V503 in the Base Study: Participants received the selected dose formulation of V503 (0.5 mL in a 3-dose regimen) from a Denmark, Norway, or Sweden site in the base study (V503-001, NCT00543543). No study vaccination will be administered in study V503-021.
  Interventions: Biological: V503
- Cohort 2: GARDASIL in the Base Study: Participants received GARDASIL (0.5 mL in a 3-dose regimen) from a Denmark, Norway, or Sweden site in the base study (V503-001, NCT00543543) and were offered the selected dose formulation of V503 (0.5 mL in a 3-dose regimen) at the conclusion of the base study. V503 vaccination was voluntary and not a condition for inclusion in Cohort 2. No study vaccination will be administered in study V503-021.
  Interventions: Biological: V503; Biological: GARDASIL

INTERVENTIONS:
Biological: V503
Biological: GARDASIL
  Groups: Cohort 2: GARDASIL in the Base Study

SUMMARY:
Protocol V503-021 is a long-term follow-up study of the V503-001 base study (NCT00543543) to evaluate the safety, immunogenicity, and long-term effectiveness of V503 vaccine in preventing cervical cancer and related precancers caused by human papillomavirus (HPV) types 16, 18, 31, 33, 45, 52, and 58. Because of the high retention of V503-001 participants from the Nordic countries, and the highly efficient screening and surveillance system there, study V503-021 will evaluate only participants from V503-001 sites in Denmark, Norway, and Sweden. The hypothesis is that V503 vaccine will remain effective for at least 30 years after the start of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Randomized into the V503-001 (NCT00543543) study from a Denmark, Norway, or Sweden site and participated in the study by receiving either the selected dose formulation of V503 or GARDASIL
* Agrees to allow passive follow-up, analysis of biopsy specimens, future contact from the National Registry Study Centers, and serum collection

Exclusion Criteria:

- There are no exclusion criteria

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants in the V503-021 long-term follow-up study received either the selected dose formulation of V503 or GARDASIL in the V503-001 (NCT00543543) base study
Sampling Method: Non-Probability Sample
Enrollment: 4453 (Estimated)
Dates: Start 2016-01-22 (Actual); Primary Completion 2040-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Combined Incidence of HPV Type 16, 18, 31, 33, 45, 52, or 58-related Cervical Intraepithelial Neoplasia (CIN) Grades 2 or 3, Adenocarcinoma In Situ (AIS), and Cervical Cancer in Cohort 1 | Up to 30 years after vaccination in V503-001 base study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Luxembourg A, Kjaer SK, Nygard M, Ellison MC, Group T, Marshall JB, Radley D, Saah A. Design of a long-term follow-up effectiveness, immunogenicity and safety study of women who received the 9-valent human papillomavirus vaccine. Contemp Clin Trials. 2017 Jan;52:54-61. doi: 10.1016/j.cct.2016.10.006. Epub 2016 Oct 21. PMID 27777126
- [Result] Kjaer SK, Nygard M, Sundstrom K, Munk C, Berger S, Dzabic M, Fridrich KE, Waldstrom M, Sorbye SW, Bautista O, Group T, Luxembourg A. Long-term effectiveness of the nine-valent human papillomavirus vaccine in Scandinavian women: interim analysis after 8 years of follow-up. Hum Vaccin Immunother. 2021 Apr 3;17(4):943-949. doi: 10.1080/21645515.2020.1839292. Epub 2020 Dec 16. PMID 33326342
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26177&tenant=MT_MSD_9011